CLINICAL TRIAL: NCT00507702
Title: Identification of Key Blood Molecular Markers for Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: Improving assay methods
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: VAR0017; 97125 (Other: Stanford University Alternate IRB Approval Number); VAR0017 (Other: Stanford University)
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Squamous Cell Carcinoma; Adenocarcinoma; Neoplasms
MeSH Terms: conditions — Carcinoma, Squamous Cell; Adenocarcinoma; Neoplasms | interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: phlebotomy — Standard of care
  Other Names: blood draw

SUMMARY:
To identify unique blood markers in cancer patients so that we can identify patients with evidence of pre-existing immunity who may be a responder to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with cancerous tumors based on biopsy or other clinical observations.
2. Patients diagnosed with non-cancerous tumors based on biopsy or other clinical observations.
3. Normal volunteers who do not have cancer or other medical conditions that may affect survival.

Exclusion Criteria:

1. Patients will be excluded if, upon clinical observation, they are under a severe septic or inflammatory condition. In these conditions, human body immune response against sepsis or inflammation should be the predominant response, and may shield or block the immune response against tumors.
2. Patients will be excluded if, upon clinical observation, they are under extremely illness situation like myocardial infarction. In such a case, the immune findings may be altered.
3. Patients will be excluded if, upon looking through their medical records, significant information required for data analysis is missing. This is because that patients' medical records will help us connect our research findings with their clinical observations, and further provide guidelines for subsequent treatment options.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumors occur predominantly in the adult population after age 30, regardless of gender and ethnic background. Therefore, our study population will consist mainly of adult subjects. We do not have any exclusion criteria based on age range, gender or ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2006-07-06 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2015-02-25 (Actual)

PRIMARY OUTCOMES:
To identify and evaluate the presence of pre-existing immunity related markers in peripheral human blood, to identify patients who may respond to IL-12 immunotherapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Norton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States